**Study Title:** Motivation Skills Training for Schizophrenia

Clinicaltrials.gov: NCT05746455

**Statistical Analysis Plan** 

Date of Approval: 12/23/2022

## **Motivation Skills Training for Schizophrenia**

We will pilot Motivation Skills Training (MST) in one outpatient mental health clinic. The goals of this study are to obtain *preliminary evidence* of target engagement (change in motivation), obtain feedback on treatment satisfaction and acceptability from service recipients and feedback from clinicians on the feasibility and clinical utility of the treatment manual. These data will inform refinement of the assessment procedures and intervention parameters. **Within-person change from pre to post MST** will be assessed using descriptive statistics and paired *t*-tests for the primary outcome, the Motivation and Pleasure Scale (**MAP**), and for the primary and secondary functional outcomes, Goal Attainment Scaling (**GAS**) and Heinrichs Carpenter Quality of Life Scale (**QLS**), respectively. However, magnitude of the effect size of improvement will be the primary focus rather than statistical significance given the small sample and pilot nature of the data. Quantitative data from a treatment satisfaction questionnaire, retention rate and rate of pre/post assessment completion will be summarized with descriptive statistics. Qualitative feedback from clinicians implementing MST will be summarized to facilitate any possible changes to procedures, training curriculum and to the treatment manual.